CLINICAL TRIAL: NCT01706458
Title: Pilot Trial of Sipuleucel-T, With or Without pTVG-HP DNA Booster Vaccine, in Patients With Castrate-Resistant, Metastatic Prostate Cancer
Brief Title: Provenge With or Without pTVG-HP DNA Booster Vaccine in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO11816; A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); NCI-2012-02026 (Registry Identifier: NCI Trial ID); 2012-0352 (Registry Identifier: Institutional Review Board)
Record Dates: First submitted 2012-10-09; First posted 2012-10-15 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
Keywords: Vaccine; pTVG-HP; Prostate Cancer; Castrate Resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T; Vaccines, DNA; regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sipuleucel-T (Active Comparator): Patients receive sipuleucel-T IV on weeks 0, 2, and 4.
  Interventions: Biological: sipuleucel-T
- sipuleucel-T with DNA Vaccine (Experimental): Patients receive sipuleucel-T as patients in arm I and pTVG-HP plasmid DNA vaccine ID on weeks 6, 8, 10, and 12, and then at 6 and 9 months.
  Interventions: Biological: sipuleucel-T; Biological: DNA Vaccine

INTERVENTIONS:
Biological: sipuleucel-T — Given IV
  Other Names: Provenge
Biological: DNA Vaccine — Given ID
  Other Names: pTVG-HP with rhGM-CSF
  Arms: sipuleucel-T with DNA Vaccine

SUMMARY:
This randomized pilot clinical trial studies sipuleucel-T with or without deoxyribonucleic acid (DNA) vaccine therapy in treating patients with prostate cancer that has not responded to previous treatment with hormones and has spread to other places in the body. Vaccines may help the body build an effective immune response to kill tumor cells. It is not yet known whether giving sipuleucel-T vaccine works better with or without DNA vaccine therapy in treating prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate)
* Metastatic disease as evidenced by the presence of soft tissue and/or bone metastases on imaging studies (computed tomography [CT] of abdomen/pelvis, bone scintigraphy)
* Castrate-resistant disease, defined as follows:

  * All patients must have received standard of care androgen deprivation treatment before trial entry (surgical castration versus gonadotropin-releasing hormone [GnRH] analogue or antagonist treatment), and subjects receiving GnRH analogue or antagonist must continue this treatment throughout the time on this study
  * Patients may have been treated previously with a nonsteroidal antiandrogen, with evidence of disease progression subsequently; subjects must be off use of anti-androgen for at least 4 weeks (for flutamide) or 6 weeks (for bicalutamide or nilutamide) prior to registration

    ** Subjects who demonstrate an anti-androgen withdrawal response, defined as a >= 25% decline in PSA within 4-6 week of stopping a nonsteroidal antiandrogen are not eligible until the PSA rises above the nadir observed after antiandrogen withdrawal
  * Castration levels of testosterone (< 50 ng/dL) within 2 weeks of registration
* Progressive disease while receiving androgen deprivation therapy defined by any one of the following as per the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) bone scan criteria or Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 during or after completing last therapy:

  * PSA: at least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, and each value >= 2.0 ng/mL
  * Measurable disease: >= 50% increase in the sum of the cross products of all measurable lesions or the development of new measurable lesions; the short axis of a target lymph node must be at least 15 mm by spiral CT to be considered a target lesion
  * Non-measurable (bone) disease: the appearance of two or more new areas of uptake on bone scan consistent with metastatic disease compared to previous imaging during castration therapy; the increased uptake of pre-existing lesions on bone scan will not be taken to constitute progression, and ambiguous results must be confirmed by other imaging modalities (e.g. X-ray, CT or magnetic resonance imaging [MRI])
* Must have >= 3 serum PSA values obtained over at least a 12 week period of time prior to registration, including the day of screening, to calculate a PSA doubling time; Note: PSA's are not required to be obtained at the same laboratory; use all PSA values that have been done in last 6 months to calculate PSA doubling time
* Life expectancy of at least 6 months
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* White blood cell >= 2000/mm^3
* Absolute neutrophil count >= 1000/mm^3
* Hemoglobin (HgB) >= 9.0 mg/dL
* Platelets >= 100,000/mm^3
* Creatinine =< 2.0 mg/dL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* Negative serology tests for human immunodeficiency virus (HIV) 1 and 2, and for active hepatitis B or hepatitis C, within 14 days of first peripheral blood collection for sipuleucel-T
* Patients must be at least 4 weeks from any prior treatments and have recovered (to < grade 2) from acute toxicity attributed to this prior treatment
* Patients must be informed of the experimental nature of the study and its potential risks, and must sign an Institutional Review Board (IRB)-approved written informed consent form indicating such an understanding

Exclusion Criteria:

* Small cell or other variant prostate cancer histology
* Patients may not be receiving other investigational agents or be receiving concurrent anticancer therapy other than androgen deprivation
* Symptomatic metastatic disease, as defined by the need for opioid analgesics for the treatment of pain attributed to a prostate cancer metastatic lesion; patients receiving opioids must receive approval from the principal investigator (PI) for eligibility
* Patients may not have been treated with prior sipuleucel-T
* Treatment with any of the following medications within 28 days of registration, or while on study, is prohibited:

  * Systemic corticosteroids (at doses over the equivalent of 1 mg prednisone daily); inhaled, intranasal or topical corticosteroids are acceptable
  * Prostate cancer (PC)-SPES
  * Saw palmetto
  * Megestrol
  * Ketoconazole
  * 5-alpha-reductase inhibitors-patients already taking 5-alpha-reductase inhibitors prior to 28 days prior to registration may stay on these agents throughout the course of therapy, but these should not be started while patients are on study
  * Diethyl stilbestrol
  * Abiraterone
  * Any other hormonal agent or supplement being used with the intent of cancer treatment
* External beam radiation therapy within 4 weeks of registration is prohibited, or anticipated need for radiation therapy (e.g. imminent pathological fracture or spinal cord compression) within 3 months of registration
* Major surgery within 4 weeks of registration is prohibited
* Prior cytotoxic chemotherapy (e.g. docetaxel, mitoxantrone, cabazitaxel) within 6 months of registration is prohibited
* Patients with a history of life-threatening autoimmune disease
* Patients who have undergone splenectomy
* Patients must not have other active malignancies other than non-melanoma skin cancers or carcinoma in situ of the bladder; subjects with a history of other cancers who have been adequately treated and have been recurrence-free for >= 3 years are eligible
* Patients with known brain metastases
* Any antibiotic therapy or evidence of infection within 1 week of registration
* Any other medical intervention or condition, which, in the opinion of the PI could compromise patient safety or adherence with the study requirements
* Patients cannot have concurrent enrollment on other phase I, II, or III investigational treatment studies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, M.D., PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Wargowski E, Johnson LE, Eickhoff JC, Delmastro L, Staab MJ, Liu G, McNeel DG. Prime-boost vaccination targeting prostatic acid phosphatase (PAP) in patients with metastatic castration-resistant prostate cancer (mCRPC) using Sipuleucel-T and a DNA vaccine. J Immunother Cancer. 2018 Mar 13;6(1):21. doi: 10.1186/s40425-018-0333-y. PMID 29534736
- See also: University of Wisconsin Carbone Cancer Center — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Started | 9 | 9
Completed | 6 | 5
Not Completed | 3 | 4
Not completed — Physician Decision | 3 | 4

BASELINE CHARACTERISTICS:
Population: Male patients, histological diagnosis of prostate adenocarcinoma and PSA recurrence following castration were eligible, provided they had evidence of metastatic disease by CT of abdomen/pelvis or bone scintigraphy. Progressive disease following last treatment required, per Prostate Cancer Working Group 2 criteria. 4 weeks from prior treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Full Range); unit: years] | 75 [67 to 82] | 72 [66 to 85] | 74 [66 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status describes a patient's level of function:
  0. is fully active, performance without restriction,
  1. is restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work,
  2. is ambulatory and capable of selfcare but unable to carry out work activities, up and about more that 50% of waking hours,
  3. is capable of limited selfcare; confined to bed or chair more than 50% of waking hours,
  4. is completely disabled; no selfcare, confined to bed or chair,
  5. is deceased
  Participants
    0 | 9 | 8 | 17
    1 | 0 | 1 | 1
Gleason score [Count of Participants; unit: Participants] — The Gleason Score is a grading system for prostate cancer severity. It is defined on a scale of 1-5 where 1 is low-grade tumor cells and 5 is high-grade tumor cells.
  Pathologists assign two Gleason grades to a biopsy; one for the predominant pattern and another for the second most predominant pattern. The two grades are added together to determine the Gleason Score (ultimately a number between 2 and 10). Scores of 2-4 tend to indicate less aggressive cancers, and 7-10 indicate more aggressive cancers.
  Participants
    < 7 | 1 | 2 | 3
    7 | 3 | 4 | 7
    8 | 0 | 2 | 2
    >/= 9 | 5 | 0 | 5
    Unknown | 0 | 1 | 1
Metastatic sites [Count of Participants; unit: Participants]
  Visceral | 2 | 0 | 2
  Bone | 2 | 5 | 7
  Distant lymph nodes | 6 | 4 | 10
Baseline PSA (ng/mL) [Median (Full Range); unit: ng/mL] | 32.6 [4.17 to 1090] | 11.2 [2.09 to 68.4] | 16.25 [2.09 to 1090]
Baseline PSA doubling time (months) [Median (Full Range); unit: months] | 2.8 [1.4 to 63.9] | 2.2 [1.0 to 25.8] | 2.55 [1.0 to 63.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immune Response Following Treatment
Description: The primary immunological goal of this study was to determine whether booster immunizations with a DNA vaccine encoding PAP could augment the number of PAP-specific effector and memory T cells following treatment with sipuleucel-T, or prolong the duration of detectable T-cell response. All subjects received a tetanus booster immunization prior to beginning the immunization series, providing a separate test of an individual's immune responsiveness. Responses to PSA, a non-target prostate specific protein, were concurrently evaluated, as were responses to GM-CSF, a component of the PA2024 fusion protein used in the preparation of sipuleucel-T.Samples were evaluated for antigen-specific IFNy or granzyme B secretion by ELISPOT, and the detection of statistically significant antigen-specific responses, that were at least 3-fold over the baseline value, and detectable more than once post-treatment, were used to define immune response to a particular antigen.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 9 | 9
Participants | 6 | 5

2. Secondary Outcome: Progression-free Survival
Description: Percentage of patients without radiographic progression at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

3. Secondary Outcome: Time to Radiographic Disease Progression
Description: Time to radiographic progression using staging obtained at month 3 as baseline for evaluation.
Time Frame: 12 months
Measure: Median (Full Range); unit: days
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 9 | 9
days | 161 [85 to 259] | 164 [85 to 343]

4. Secondary Outcome: Measure Prostate-specific Antigen (PSA) Doubling Time
Description: PSA doubling times were calculated from PSA values obtained up to 6 months from day 1 of study treatment. An increase in the PSA doubling time to at least double the baseline value will be defined as a PSA doubling time "response".
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 9 | 9
months | 2.5 [1.1 to 8.8] | 2.6 [1.7 to 3.6]

5. Other Pre Specified Outcome: Overall Survival: Median Time to Death From Any Cause
Description: Overall survival is defined as the time interval from randomization to death from any cause or to the last follow-up in censored patients.
Time Frame: up to approximately 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 9 | 9
months | 32.3 [7.7 to 66.7] | 29.6 [14.6 to 46.0]
Statistical Analysis 1: Comparison: Sipuleucel-T vs Sipuleucel-T With DNA Vaccine; Test type: Other; p = 0.9060, Log Rank

6. Other Pre Specified Outcome: Number of Circulating Tumor Cells
Time Frame: 6 months
Population: This outcome measure was not determined because there was no progression free survival at one-year.
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: PAP-specific Antibody and T-cell Immune Responses Following Treatment With Sipuleucel-T and DNA Vaccine
Description: A response resulting from immunization was defined as a PAP-specific response detectable more than once post-treatment that was both significant (compared to media only control), at least 3-fold higher than the pre-treatment value, and with a frequency> 1:100,000 PBMC. An antibody response was defined as any increase in titer over baseline.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 9 | 9
Participants
  Interferon Gamma Response | 3 | 2
  Granzyme B | 4 | 4
  Antibody Response | 3 | 5

8. Other Pre Specified Outcome: Logistic Regression Analysis Will be Conducted to Evaluate Whether PAP-specific Immune Response is Associated With Prolonged (1-year) Progression-free Survival.
Description: Not performed because no progression free survival at one year.
Time Frame: 12 months
Population: This outcome measure was not determined because there was no progression free survival at one-year.
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Logistic Regression Analysis Will be Conducted to Evaluate Whether Baseline Immune Responses Predict for Immune Responses Elicited/Augmented Following Treatment With Sipuleucel-T +/- DNA Vaccine.
Description: Not performed because no progression free survival at one year.
Time Frame: 12 months
Population: This outcome measure was not determined because there was no progression-free survival at one-year.
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: The Detection of Antigen Spread to Other Prostate Associated Antigens, and the Identification of Specific Antigens Recognized, Will be Analyzed Descriptively.
Description: Not performed because no progression free survival at one year.
Time Frame: 12 months
Population: This outcome measure was not determined because there was no progression free survival at one-year.
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Overall, patients were followed for a mean of 24 months.
Arm/Group | Sipuleucel-T | Sipuleucel-T With DNA Vaccine
All-Cause Mortality (participants affected / at risk) | 5/9 | 8/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=9) | Sipuleucel-T With DNA Vaccine (N=9)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=9) | Sipuleucel-T With DNA Vaccine (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (5)
Fever (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 4 (6)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (3)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Heahache (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT01706458/Prot_SAP_000.pdf